CLINICAL TRIAL: NCT07185191
Title: A Pre-market Randomized Clinical Trial to Evaluate the Safety and Clinical, Functional and Aesthetic Benefits of Polynucleotide (PN HPT™) Infiltration in the Treatment of Interdental Papilla and Marginal Soft Tissue Deficits
Brief Title: Evaluation of the Safety and Performance of the Medical Device RDM36 in the Treatment of Periodontal Gingival Contraction and in Black Triangles Syndrome (BTS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mastelli S.r.l (Industry)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHAPE STUDY
Record Dates: First submitted 2025-08-06; First posted 2025-09-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Black Triangles Syndrome (BTS); Periodontal Gingival Contraction
Keywords: BTS; Polynucleotides; Black Triangles Syndrome; PN HPT; Papilla; Tissue deficits; gingival contraction; Periodontal
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (RDM36) (Experimental)
  Interventions: Device: RDM36
- Control group (Sham Comparator)
  Interventions: Drug: Saline Solution (NaCl 0,9%)

INTERVENTIONS:
Device: RDM36 — Patients treated with RDM36; two perpendicular infiltrations (buccal, palatal) of a quantity of 0.2 ml of PN HPT
  Arms: Treatment group (RDM36)
Drug: Saline Solution (NaCl 0,9%) — patients treated with saline solution; two perpendicular infiltrations (buccal, palatal) of a quantity of 0.2 ml of saline solution
  Arms: Control group

SUMMARY:
The treatment of black triangles in modern dentistry involves various approaches, both surgical and nonsurgical. Surgical methods aim to reconstruct or preserve gingival tissue using techniques such as soft tissue flaps or augmentation. Some invasive surgical methods proposed for papilla reconstruction and correction of black triangle recession include repeated interproximal curettage, Beagle's pedicle graft procedure, free epithelialized and de-epithelialized gingival grafts, and subepithelial connective tissue grafts. The success rate of surgical augmentation depends on the thickness of the gingiva biotype. Orthodontic treatment can also be used to reshape and decrease the embrasure space.

An alternative option is minimally invasive procedures for tissue re-volumizing and papilla anatomical-functional reconstruction. Hyaluronic acid (HA) has been used for minimally invasive papilla reconstruction, leveraging its volumizing filler effect.

Non-surgical strategies based on hyaluronan are gaining ground internationally. The immediate goal of minimally invasive treatment for interdental papilla loss and black triangle disease is mechanical protection and gingival restoration. Promoting tissue hydration, fibroblast vitality, and collagen deposition may offer a long-term regenerative medicine solution. Additionally, natural-origin, High Purification Technology Polynucleotides (PN HPTTM) are exploited for wound healing and counteracting connective tissue depletion.

PNs-based medical devices are widely used in Europe and other countries for various indications, including orthopedics (intra-articular administration), dermatology (intra-dermal injections), and vulvo-vaginal application.

PNs have minimal protein contaminants and allergic risks due to advanced purification techniques. Their hydrophilic nature provides hydration and acts as a volume enhancer. Recent in vitro studies demonstrate improved gingival fibroblast viability and collagen deposition with PNs.

The purpose of this clinical investigation is to assess the safety and clinical performance of RDM36 in the treatment of periodontal gingival contraction and in black triangles syndrome (BTS).

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide written informed consent (ICF) for the study.
2. Males and females.
3. Be aged 18 years or older at the time of signing the informed consent.
4. Subjects have to show at least one anterior interdental papilla recession in the smile zone according to Jemt's classification (BTS).
5. The teeth near the interdental papilla recession must have the contact point.
6. Absence of periodontal diseases.
7. Subjects with adequate knowledge of domiciliary oral hygiene practices, as measured by the following parameters: FMPS (full mouth plaque score) and FMBS (full mouth bleeding score) values <10%.
8. Absence of plaque and bleeding on probing at the site of interest.
9. Absence of retentive factors at the site of interest.

Exclusion Criteria:

1. Subjects with active periodontitis.
2. Presence of an acute infection in the oral cavity or upper respiratory tract.
3. Pregnancy or breastfeeding or planning to conceive from the clinical evaluation for enrollment up to 120 days after the end of the treatment.
4. Subjects must not be Smokers more than 10 cigarettes per day.
5. Presence of bleeding disorders or taking medications that affect blood clotting (e.g., coumarin-type drugs or platelet aggregation inhibitors).
6. Presence of systemic diseases that could affect periodontal health.
7. Patients with autoimmune diseases.
8. Known or suspected allergy to seafood products.
9. Psychiatric or behavioral disorders or substance abuse that would interfere with the necessary cooperation for the study.
10. Presence of infra-bony defects associated with pocket or papilla contraction and visible on X-ray as well as detectable on probing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse device effects (ADE) and serious adverse device effects (SADE) - Safety outcome | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
Clinical performance of RDM36 in the 2D modification of the "black triangle" lesion through photographic documentation using Image-J software obtained from a scan (TRIOS 6 3Shape intraoral scanner) and from superimposition compared to baseline | Visit 2 (6 ± 1 weeks)

SECONDARY OUTCOMES:
Clinical performance of RDM36 in the 2D modification of the "black triangle" lesion through photographic documentation using Image-J software obtained from a scan (TRIOS 6 3Shape intraoral scanner) and from superimposition compared to baseline | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
Patients' subjective evaluation of the aesthetic improvement of black triangle syndrome through the Visual Analogue Scale (VAS, 0-10 score, where 0=very satisfactory and 10=unsatisfactory) | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
Patients' subjective evaluation of the aesthetic improvement of black triangle syndrome through the Global Aesthetic Improvement Scale (GAIS) | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
  GAIS, rated on a 5-point scale (1= very much/extremely improved; 2= much improved; 3= improved; 4= no change; 5= worse)
Patients' subjective evaluation of the aesthetic improvement of black triangle syndrome through the Likert scale | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
  5 point-Likert scale, from 1 to 5 indicating how satisfied is the patient (1 - Extremely dissatisfied, 5 - Extremely satisfied)
Evaluation of the clinical performance of RDM36 in the 3D modification of the "black triangle" lesion through a scanner volumetric analysis (TRIOS 6 3Shape) and Blender software. | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
Papilla's colorimetric evaluation using a colorimeter (OPTISHADE STYLEITALIANO) that will objectively rank the stability or improvement of gingival health on a red scale | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
Periodontal health evaluation through Plaque Index (PI) | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
  The PI is a dichotomous parameters (0 = absence, 1 = presence)
Periodontal health evaluation through Bleeding on Probing (BOP) | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
  The BOP is a dichotomous parameters (0 = absence, 1 = presence)
Periodontal health evaluation through Recession (REC) at the study site | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
  REC is measured in millimeters (PD: < 4 mm = health, > 4mm = periodontal disease)
Periodontal health evaluation through Probing Depth (PD) at the study site | From enrollment to the end of treatment at 26 weeks (± 2 weeks) from baseline
  PD is measured in millimeters (PD: < 4 mm = health, > 4mm = periodontal disease)

IPD SHARING:
Plan to Share IPD: Undecided